CLINICAL TRIAL: NCT00821808
Title: A Phase I, Randomized, Open-label, One-arm, Active Controlled Study to Evaluate the Pressure Interface Between Device and Skin of a Compression Device and Profore® on Healthy Volunteers
Brief Title: A Pressure Relted Study Comparing a Compression Device and Profore® on Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CW-0500-08-U347
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Compression Device — The compression device will be worn for 8 hours each day on one leg. The device will be applied by the same clinician every morning.Interface pressure measurements will be made in both the sitting and standing position at three locations on the leg at the following time intervals:
  * Immediately following device application
  * 1 hour
  * 4 hours
  * 8 hours
Device: Profore® — Profore® will be worn for 8 hours each day on opposite leg. Profore® will be applied by the same clinician every morning.Interface pressure measurements will be made in both the sitting and standing position at three locations on the leg at the following time intervals:
  * Immediately following device application
  * 1 hour
  * 4 hours
  * 8 hours

SUMMARY:
This phase I Healthy Volunteer study will evaluate the pressure interface between the devices (a compression device and Profore®) and the skin, using the PicoPress(TM) pressure transducer at specified time intervals in three distinct locations on the leg, in both the sitting and standing position. It will also assess the variability of interface pressure following application under each test device for each subject over a period of three days (three separate applications).

ELIGIBILITY:
Inclusion Criteria:

* over 18 years, willing and able to provide written informed consent.
* able to wear the compression device and Profore® and follow the requirements of the clinical investigation plan
* an ankle to brachial pressure index (ABPI) of 0.9 or greater
* CEAP classification C0-C2
* healthy volunteers

Exclusion Criteria:

* history of skin sensitivity to any of the components of the study product
* participated in a previous clinical study within the past 3 months
* active Deep Vein Thrombosis (DVT) or a recent DVT within the last 3 months
* exhibited any other medical condition which, according to the Investigator, justifies the subject's exclusion from the study
* leg sizes outside the following range:

  * Ankle - 12cm to 44cm
  * Calf - 22cm to 60cm
  * Below knee - 22cm to 68cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the amount of pressure and the variability of interface pressure of the two devices on application | 3 days
To evaluate pressure change of the interface pressure with the compression device and Profore® over time | 3 days
Safety will be evaluated by the nature and frequency of adverse events. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Vanscheidt, MD, Principal Investigator — Hautarzt Phlebologe Allergologe
Locations (1):
- Hautarzt Phlebologe Allergologe, Freiburg im Breisgau, Germany